CLINICAL TRIAL: NCT06663865
Title: Investigating the Effects of Dairy Phospholipids on Sleep and Daytime Function in Healthy Adults.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 66CH3
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-09

CONDITIONS: Sleep; Morning Alertness; Evening Alertness; Diurnal Cortisol
Keywords: Sleep; Daytime function; diurnal cortisol; Morning alertness; Evening alertness; dreams
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo-controlled, parallel groups design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Treatment will be blinded according to the randomisation schedule by a research who has no other involvement in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bioactive whey protein concentrate containing dairy phospholipids (Experimental): 40g pre weighed powder to be mixed with 350ml of water. Consumed one daily for 12 weeks alongside their fattiest meal of the day.
  Interventions: Dietary Supplement: Active
- Placebo Powder (Placebo Comparator): Placebo powder matched for macro-nutrient and caloric content containing pea protein around 40g powder mixed with 350ml of water consumed once daily for 12 weeks alongside fattiest meal of the day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Active — 40g bio-active whey protein concentrate powder containing dairy phospholipids
  Other Names:
  Active Treatment
  Arms: Bioactive whey protein concentrate containing dairy phospholipids
Dietary Supplement: Placebo — Around 40g pea protein powder not containing dairy phospholipids
  Other Names:
  Placebo Treatment
  Arms: Placebo Powder

SUMMARY:
The aim of the study is to investigate the effects of 6- and 12- week supplementation of a bioactive whey protein concentrate drink containing dairy phospholipids on sleep and daytime function parameters in healthy adults.

The proposed randomised, double-blind, placebo-controlled parallel groups design methodology will assess the sleep and daytime function effects (both self-reported and physiological) of 40g per day of bioactive whey protein concentrate in the form of a powder that the participant will be required to mix with 350ml of water and matched placebo prior to (baseline) and after -6 week and -12 week supplementation. The trial will utilise actigraphy sleep watches and online cognitive assessments alongside saliva sampling, sleep diaries, and self-report questionnaires as measures of the outcome variables.

70 participants will participate, aged 25-49, and self-reported as being in good health. Participants will be supplied with either the active treatment or the placebo (allocated by a randomised schedule) whilst visiting the research centre for the testing appointments and will take treatment home to consume daily for the duration of the study. Participants will record time of taking treatment each day in a treatment diary which will be returned to the research centre, along with any unused treatment, upon completion of the study.

DETAILED DESCRIPTION:
The study will follow a randomised, placebo-controlled, double-blind, parallel groups design. Participants will be given 12-weeks; worth of either placebo or active treatment to be consumed at home each day (double blinded), will attend all 7 appointments required at the research centre, will complete the at home treatment diary daily, as well as completing the at home tasks.

Participants will attend the research centre on six separate occasions, which will include a screening/training visit, pre intervention testing visit, a mid-point testing visit (at 6 weeks), a completion of intervention testing visit (at 12 weeks), as well as 2 collection visits to retrieve equipment for the at home tasks. 7 Appointments in total including the online appointment to check for eligibility. The remote screening session will be completed via telephone call and will comprise briefing on the requirements for the study, answering any initial questions, obtaining of informed consent via completion of an online consent form, health screening, collection of demographic information, and completion of the Caffeine Consumption Questionnaire (CCQ).

The introductory/training visit to the laboratory will begin with physiological eligibility measures that cannot be completed remotely (e.g., blood pressure, height and weight, waist-to-hip ratio) followed by training on the cognitive and mood measures. Instructions on the at home tasks will also be given here including how to provide saliva samples, how to access and use Cognimapp (at home cognitive assessment tool), and how to use the actigraphy sleep watches.

The study will include 70 healthy participants aged between 25-49 years, who will receive 12 weeks; worth of either 40g per day of bioactive whey protein concentrate powder containing dairy phospholipids (to be mixed with 350ml of water to form a drink), or a similar of placebo powder. Participants will be randomly allocated to either the treatment or placebo group and neither the participant nor the researcher will know which group they have been allocated to. Full instructions of how and when to take treatment each day will be explained to the participants when treatment is given at testing visit 1.

On each of the three study days (Day 1, 42, and 84) participants will attend the research centre, having abstained from alcohol for 24 hours, and caffeine overnight, following a standardised breakfast of cereal and/or toast at home no later than 1 hour prior to arrival. After completing the cognition tasks outlined in a separate protocol, The participants will be administered their treatment and instructed on/reminded of how it should be taken each day (Day 1 and 42). Participants will be asked to return any unused treatment at visit 2 and 3, along with their treatment diary. Participants will additionally complete a treatment guess form at their final visit and will be fully debriefed.

Participants will need to attend the research centre 7 days prior to each of the testing visits (this will be the training visit in the case of Day 1 testing visit), to retrieve their at home testing equipment. This will include an actigraphy sleep watch, a saliva sampling kit, and instructions on how to provide a saliva sample, how to use the actigraphy sleep watches, and how to access the online cognitive assessments. They will also be provided with a sleep diary.

Participants will wear the sleep watches for 7 days prior to each of the 3 testing visits. They will also complete a sleep diary for this duration. In addition, participants will provide saliva samples at 4 different time points (wakening, 30 minutes post wake, 45 minutes post wake, before bed) for 3 consecutive days before each testing visit. Finally, participants will also complete several cognitive tasks for 3 consecutive mornings and evenings before each testing visit. They will access the cognitive tasks through a online software (Cognimapp) that allows participants to complete cognitive assessments from home. The assessments will be measures of morning and evening alertness and will also include a alertness visual analogue scale.

As outlined in another protocol, participants will also be completing a battery of questionnaires the day before the testing visits. Within this battery of questionnaires, they will also complete a dream questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Participants must self-assess themselves as being in good health.
* Participants must be aged 25 to 49 years at the time of giving consent.
* Participants must be a native speaker of English or fluent in English

Exclusion Criteria:

* Have any pre-existing medical conditions/illness which will impact taking part in the study. There may be other, unforeseen exceptions and these will be considered on a case-by-case basis: i.e., participants may be allowed to progress to screening if they have a condition/illness which would not interact with the active treatments or impede performance. It is therefore worth discussing any medical conditions with the researcher prior to booking appointments
* Are currently taking any prescription medications (NOTE the explicit exceptions to this are contraceptive treatments for female participants, and those taking "as needed" in the treatment of asthma and/or hay fever. There may be other instances of medication use which, where no interaction with the active treatment is likely, and which would not be expected to have any impact on brain function, participants may be able to progress to screening
* Have high blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg). NOTE: that we must measure this in the lab using our blood pressure monitors and can only use our measurements to assess eligibility rather than home or GP readings
* Have a Body Mass Index (BMI) outside of the range 18.5-35 kg/m2.
* Are pregnant, seeking to become pregnant or lactating.
* Have learning and/or behavioural difficulties such as dyslexia or ADHD.
* Have a visual impairment that cannot be corrected with glasses or contact lenses (including colour-blindness)
* Smoke tobacco or vape nicotine or use nicotine replacement products (if you have recently quit smoking or using replacements you must have stopped using them altogether for a period of 3 months before participating in this study)
* Have excessive caffeine intake (500 mg per day). Note: This will be calculated at screening but feel free to query this with the researcher prior to attendance
* Have relevant food allergies/ intolerance/ sensitivities
* Have taken antibiotics within the past 4 weeks.
* Have taken dietary supplements e.g., vitamins, omega 3 fish oils etc. in the last 4 weeks (Note: participation is possible following a 4 week supplement wash out prior to participating and for the duration of the study on the proviso that the supplements they are taking are out of choice and not medically prescribed or advised. Please discuss with the researcher if unsure. NOTE: we would never advise stopping supplements prescribed by your doctor e.g., iron, calcium etc., only those you use out of choice)
* Have any health condition that would prevent fulfilment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken)
* Are unable to complete all of the study assessments (this will be assessed by the researcher at the training appointment)
* Are currently participating in other clinical or nutrition intervention studies, or have in the past 4 weeks
* Have been diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months.
* Have been diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months, including a medical diagnosis of anxiety or depression.
* Suffers from frequent migraines that require medication (more than or equal to 1 per month)
* Have any sleep disorders or take any sleep medications.
* Routinely work night shifts
* Have any known active infections.
* Does not have a bank account (required for payment)
* Are non-compliant with regards treatment consumption
* Follow an "extreme" or very "strict" diet i.e., Keto, very high protein, sugar free, raw paleo etc.
* Are planning a major lifestyle change regarding diet or exercise regime in the next 3 months.
* Experienced an event (professional or personal) that is likely to have impacted your emotional and/or psychological state within the last 8-10 weeks (for example but not restricted to change of professional function, death of a family member, divorce, surgery, accident etc)
* Have an upcoming event (personal or professional) that is likely to affect your emotional, psychological state or hormonal state planned during the next 8-10 weeks, including but not limited to job change, house move, important medical exam etc.
* Have any oral disease such as gingivitis
* Are planning any overseas travel with significant time zone differences

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10-28 (Estimated); Primary Completion 2025-06-27 (Estimated); Study Completion 2025-06-27 (Estimated)

PRIMARY OUTCOMES:
Sleep quality - Objective sleep quality measured through actigraphy sleep watches | prior to (baseline) and following chronic dose of intervention at 6 weeks and 12 weeks.
  Average scores across 7 days. Scores for sleep onset, total sleep time, wake after sleep onset, awakenings, average awakening, and efficiency of sleep will be averaged

SECONDARY OUTCOMES:
Acute self-reported state anxiety via the Anticipated Versus Experienced Demand Questionnaire | prior to (baseline) and following 6- and 12-week chronic intervention
  Completed morning and evening for 3 consecutive days at each time point (baseline, following 6- and 12-week intervention). Self-report 12 item measure related to state anxiety. 4-point scale with the following options; "not at all", "Somewhat", "Moderately", and "Very much".
Cognitive and somatic anxiety via the Anticipated Versus Experienced Demand Questionnaire | prior to (baseline) and following 6- and 12-week chronic intervention
  Completed morning and evening for 3 consecutive days at each time point (baseline, following 6- and 12-week intervention). Self-report 27 item measure related to cognitive and somatic anxiety. 4-point scale with the following options; "Not at all", "Somewhat", "Moderately", and "Very much".
Anticipated and Experienced Demand via the Anticipated Versus Experienced Demand Questionnaire | prior to (baseline) and following 6- and 12-week chronic intervention
  Completed morning and evening for 3 consecutive days at each time point (baseline, following 6- and 12-week intervention). Self-report 5 item scale completed morning and evening to measure anticipated (morning) versus experienced (evening) demand of the day.
Perceived Stress via the Perceived Stress Scale: | prior to (baseline) and following 6- and 12-week chronic intervention
  10-item measure, summed to create a single value with higher scores indicating higher levels of stress.
Depression, Anxiety and Stress Scale (DASS-21) | Prior to (baseline) and following 6- and 12-week chronic intervention
  21 item measure, summed to create 3 component scores; depression, anxiety, and stress.
Fatigue Assessment Scale (FAS) | prior to (baseline) and following 6- and 12-week chronic intervention
  10-item measure, summed to create a measure of over perceived fatigue.
Perceived Stress Reactivity Scale (PSRS) | prior to (baseline) and following 6- and 12-week chronic intervention
  23-item measure, summed to create measures of prolonged reactivity, reactivity to work overload, reactivity to social conflict, reactivity to failure, reactivity to social evaluation, and perceived stress reactivity.
The Cohen-Hoberman Inventory of Physical Symptoms (CHIPS) | prior to (baseline) and following 6- and 12-week chronic intervention
  33-item measure, summed to create a measure of number of health complaints in the previous 2 weeks.
Self-reported morning alertness via visual analogue scale (VAS) | prior to (baseline) and following 6- and 12-week chronic intervention
  Digital visual analogue scale completed each morning for 3 consecutive days at each of the 3 time points (baseline, following 6-, and 12- week supplementation). 21x100mm line anchored at either end by "Alter" and "inattentive".
Self-reported evening alertness via visual analogue scale (VAS) | prior to (baseline) and following 6- and 12-week chronic intervention
  Digital visual analogue scale completed each evening for 3 consecutive days at each of the 3 time points (baseline, following 6-, and 12- week supplementation). 21x100mm line anchored at either end by "Alter" and "inattentive".
Diurnal cortisol measured through saliva sampling | prior to (baseline) and following 6- and 12-week chronic intervention
  Diurnal cortisol levels measured via morning (X3) and evening (X1) saliva samples for three consecutive days at each time point (baseline, following -6 and 12- week supplementation).
Subjective sleep via the Patient-Reported Outcome Measurement, Information System Sleep Disturbance Scale- short form (PROMIS-SD) | prior to (baseline) and following 6- and 12-week chronic intervention
  8-item measure, summed to create a single value with higher scores indicating higher levels of sleep disturbances.
Objective morning alertness via the Choice Reaction Time (CRT) task | prior to (baseline) and following 6- and 12-week chronic intervention
  Cognition task completed on smartphones via an online cognition website "cognimapp" sent to participant via a link from the researcher for 3 consecutive mornings at each of the 3 time points (baseline, following 6-, and 12- week supplementation). Includes 50 stimuli and scored for percentage of correct responses and reaction time (msec).
Objective morning alertness via the Digit Vigilance (DV) task | prior to (baseline) and following 6- and 12-week chronic intervention
  Cognition task completed on smartphones via an online cognition website "cognimapp" sent to participant via a link from the researcher for 3 consecutive mornings at each of the 3 time points (baseline, following 6-, and 12- week supplementation). Outcomes include accuracy, mean reaction time and number of false alarms.
Objective morning alertness via the Peg and Ball task | prior to (baseline) and following 6- and 12-week chronic intervention
  Cognition task completed on smartphones via an online cognition website "cognimapp" sent to participant via a link from the researcher for 3 consecutive mornings at each of the 3 time points (baseline, following 6-, and 12- week supplementation). Task outcomes include average thinking time, completion time and errors.
Objective Evening alertness via the Choice Reaction Time (CRT) task | prior to (baseline) and following 6- and 12-week chronic intervention
  Cognition task completed on smartphones via an online cognition website "cognimapp" sent to participant via a link from the researcher for 3 consecutive evenings at each of the 3 time points (baseline, following 6-, and 12- week supplementation). Includes 50 stimuli and scored for percentage of correct responses and reaction time (msec).
Objective evening alertness via the Digit Vigilance (DV) task | prior to (baseline) and following 6- and 12-week chronic intervention
  Cognition task completed on smartphones via an online cognition website "cognimapp" sent to participant via a link from the researcher for 3 consecutive evenings at each of the 3 time points (baseline, following 6-, and 12- week supplementation). Outcomes include accuracy, mean reaction time and number of false alarms.
Objective evening alertness via the Peg and Ball task | prior to (baseline) and following 6- and 12-week chronic intervention
  Cognition task completed on smartphones via an online cognition website "cognimapp" sent to participant via a link from the researcher for 3 consecutive evenings at each of the 3 time points (baseline, following 6-, and 12- week supplementation). Task outcomes include average thinking time, completion time and errors.

OTHER OUTCOMES:
Exploratory outcome: Changes to dream recall | prior to (baseline) and following 6- and 12-week chronic intervention
  Measurement of multiple aspects of dreaming including frequency, type, intensity, and attitudes/emotions towards dreams. Measured at 3 time points; baseline, following 6 weeks supplementation, and following 12 week supplementation.

IPD SHARING:
Plan to Share IPD: No